CLINICAL TRIAL: NCT00002970
Title: A Phase II Study of Compound 506U78 in Patients With Refractory T-Cell Malignancies-POG/CCG Intergroup Study
Brief Title: 506U78 in Treating Patients With Refractory Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01836; P9673; CCG-P9673; POG-9673; CDR0000065478; U10CA098543 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-08-11 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Lymphoblastic Lymphoma; T-cell Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nelarabine; Methotrexate; merphos; Cytarabine; Hydrocortisone

ARMS (1):
- Arm I (Experimental): GROUP 1: Patients receive a 1 hour infusion of compound 506U78 daily for 5 days in the absence of neurologic toxicity. The course repeats every 21 days. If a first relapse T-cell ALL study of higher priority is not open, then the patient may continue to receive the drug every 21 days for a maximum of 2 years provided that the patient has achieved a second complete response.
  GROUPS 2 and 4: Patients receive compound 506U78 every 21 days for a maximum of 2 years, in the absence of disease progression. After 3 courses a patient may be given CNS prophylaxis with triple intrathecal therapy (TIT), consisting of methotrexate, cytarabine and hydrocortisone after consultation with study coordinator. TIT should be given every 12 weeks.
  GROUP 3: Patients receive compound 506U78 every 21 days for a maximum of 2 years, in the absence of disease progression. TIT will be given on day 1 of weeks 1-4, 6, 9 and every 6 weeks for 12 weeks, and then every 9 weeks thereafter. This stratum is open.
  Interventions: Drug: nelarabine; Drug: methotrexate; Drug: cytarabine; Drug: therapeutic hydrocortisone

INTERVENTIONS:
Drug: nelarabine — Given IV
  Other Names: 506U78; Arranon; GW506U78
Drug: methotrexate — Given IT
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: cytarabine — Given IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: therapeutic hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Cetacort; Cort-Dome; Cortef

SUMMARY:
Phase II trial to study the effectiveness of 506U78 in treating patients with recurrent or refractory hematologic cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate to compound 506U78 (2-amino-9-b-D-arabinofuranosyl-6-methoxy-9H-purine) administered as a 1 hour infusion daily for 5 days in patients with recurrent T-cell malignancies.

II. Determine the toxicities of compound 506U78 in this group of patients. III. Correlate the biochemical pharmacology of compound 506U78 (e.g., ara-G nucleotides in leukemic blasts and CSF concentrations) with clinical response.

IV. Determine the impact of compound 506U78 therapy on survival and duration of response of patients with recurrent T-cell malignancies.

OUTLINE: Patients are stratified according to disease characteristics: Group 1: T-cell ALL or NHL in first relapse (greater than 25% bone marrow blasts, with or without concomitant extramedullary relapse other than CNS); Group 2: T-cell ALL or NHL in second or later relapse (greater than 25% bone marrow blasts, with or without concomitant extramedullary relapse other than CNS); Group 3: T-cell ALL or NHL with positive bone marrow and CSF (greater than 5% bone marrow blasts and CNS 2 or 3 involvement); Group 4: Extramedullary relapse and less than 25% blasts in the bone marrow (excluding isolated CNS relapse)

GROUP 1: Patients receive a 1 hour infusion of compound 506U78 daily for 5 days in the absence of neurologic toxicity. The course repeats every 21 days. If a first relapse T-cell ALL study of higher priority is not open, then the patient may continue to receive the drug every 21 days for a maximum of 2 years provided that the patient has achieved a second complete response.

GROUPS 2 and 4: Patients receive compound 506U78 every 21 days for a maximum of 2 years, in the absence of disease progression. After 3 courses a patient may be given CNS prophylaxis with triple intrathecal therapy (TIT), consisting of methotrexate, cytarabine and hydrocortisone after consultation with study coordinator. TIT should be given every 12 weeks.

GROUP 3: Patients receive compound 506U78 every 21 days for a maximum of 2 years, in the absence of disease progression. TIT will be given on day 1 of weeks 1-4, 6, 9 and every 6 weeks for 12 weeks, and then every 9 weeks thereafter. This stratum is open.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or recurrent acute lymphocytic leukemia (ALL) or non-Hodgkin's lymphoma (NHL) with bone marrow involvement (T-cell disease only)
* Isolated CNS relapse not eligible
* Performance status - Karnofsky 50-100%
* At least 8 weeks
* Bilirubin no greater than 1.5 mg/dL
* SGPT less than 5 times normal
* Creatinine normal for age
* Creatinine clearance or GFR at least 60 mL/min/1.73m2
* No severe uncontrolled infection
* No concurrent biologic therapy
* Recovered from toxic effects
* At least 6 weeks from administration of nitrosoureas
* No concurrent endocrine therapy
* At least 6 weeks from administration of craniospinal or hemi pelvic radiotherapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 1997-06; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Early marrow CR plus PR rate at day 21 | Day 21
  CR is defined by an M1 marrow which requires blast counts below 5%. PR is defined by an M2 marrow which requires blast counts below 25%.

SECONDARY OUTCOMES:
Remission duration | Up to 2 years
6 month cumulative event-free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Berg, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States